CLINICAL TRIAL: NCT02639117
Title: Photodynamic Therapy and Vismodegib for Multiple Basal Cell Carcinomas
Acronym: PDT-Vismo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1511201549
Record Dates: First submitted 2015-12-14; First posted 2015-12-24 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Basal Cell Carcinoma
Keywords: basal cell carcinoma, photodynamic therapy, vismodegib
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vismodegib (Other): Vismodegib 150 mgs po qd. Open label.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — Vismodegib 150 mgs po qd for 3 months
  Other Names: Erivedge

SUMMARY:
This is a Phase 1 single site study to evaluate the safety and efficacy of a combination therapy that includes the administration of vismodegib and photodynamic therapy (PDT) using aminolevulinic acid (20 percent ALA) for multiple basal cell carcinomas. All subjects will receive vismodegib 150mg by mouth every day for 3 months, and undergo three PDT sessions with topical application of ALA. The PDT will be first administered at 7+ 4 business days after the beginning of the Erivedge and at 45 + 5 business days and then at 90 + 10 business days.

Primary Objective The primary objective of this study is to determine the safety of photodynamic therapy (PDT) with vismodegib (combination therapy) for patients with multiple BCC.

3.2 Secondary Objective To evaluate the overall response rate (ORR) to the combination therapy in patients with multiple BCCs.ORR is defined as the proportion of evaluable study subjects who has complete or partial response to the study treatment.

DETAILED DESCRIPTION:
Use of PDT for the treatment of BCC Indications for PDT include superficial and nodular BCC. Eight randomized clinical trials have reported the results of PDT for superficial or nodular BCC with a total of 1583 patients. Results of the meta analysis showed overall complete clearance of PDT was 86.4 % compared to 98.2 % for surgery. The 1 year recurrence for PDT was 10.3 % vs 0. 6% for surgery. Cosmetic outcomes were much better with PDT than surgery. (Wang, 2015).

A randomized controlled trial of PDT with MAL versus surgical excision in 196 patients with superficial BCC showed a 9.3% recurrence rate for PDT versus a 0% recurrence rate for surgery at 12 months. However, the good-to-excellent cosmetic outcome was 94% and 60% for patients treated with PDT and surgical excision, respectively. Similarly, in trials of PDT versus surgery for nodular BCC, recurrence rates are less than 5% for surgery versus 14% to 30% for PDT with ALA. As with superficial BCC, cosmetic effects are consistently shown to be more favorable with PDT with ALA (Wang, 2015). In the largest single institution experience with 1440 nodular and superficial BCCs, PDT using systemically administered porfimer sodium showed an initial (6-month) complete response rate of 92%, with a recurrence rate of less than 10% at 4 years. At this same institution, a 92% complete response rate was achieved with PDT with topical ALA in 330 patients with superficial BCC, but the response rate dropped to 71% in 75 patients with nodular BCC.

In a multicenter randomized trial of PDT with MAL versus cryotherapy for superficial BCC, complete response rates at 3 months were 97% and 95%, respectively, with 5-year recurrence rates of 22% and 20% for PDT with MAL and cryotherapy, respectively. In this study, the excellent-to-good cosmetic outcome was 89% for PDT with MAL and 50% for cryotherapy.

Several clinical studies have reported an increase in the initial response rate with a lower recurrence rate after repeated PDT sessions. Initial responses usually are apparent between 3-6 months after treatment when the skin has healed over and treatment related changes have resolved. Cycles of MAL PDT repeated after 3 months for persistent BCC has been shown to offer high and durable response rates. Both efficacy and safety have also been demonstrated using repeated sessions with red or blue light at follow up times of 3, 6 and 12 months. At Roswell Park Cancer Institute, Oseroff and colleagues safely used repeated sessions of ALA PDT in children with BCNS (multiple BCC), and Gilchrest also reported the benefits of ALA PDT with red light at 2-4 month interval treatments.

The most common adverse event with either ALA or MAL PDT is the burning or stinging pain experienced by patients during illumination. Zeitouni and colleagues published their retrospective and prospective data using a 2 step irradiance approach with ALA/MAL PDT and red light in non BCNS patients with multiple BCC. Follow up times ranged from 6-24 months. The 2 step irradiance schedule (bilevel) effectively minimized the treatment related pain and maintained good clinical outcomes (Zeitouni x 2).

ELIGIBILITY:
Inclusion Criteria

Patients will be included in the study based on the following criteria:

* Male or non-childbearing potential females, at least 18 years of age (Female patients who meet at least one of the following criteria are defined as women of non-childbearing potential)
* ≥ 50 years old and naturally amenorrheic for ≥ 1 year
* Permanent premature ovarian failure confirmed by specialist gynecologist
* Previous bilateral salpingo-oophorectomy or hysterectomy
* XY karyotype, Turner's syndrome, or uterine agenesis
* Diagnosis of BCC with at least 4 nodular lesions that measure 0.5 cm to 5 cm in diameter, located on the head and neck, trunk or extremities.
* Diagnosis must be confirmed clinically at baseline with 1-2 lesions having been biopsied no sooner than 2 weeks prior to treatment.
* Patients who may have high burden of disease ie large lesions, who are non-surgical candidates or who refuse surgery.
* Non-surgical candidates, who may be able to undergo resection of selected single, individual lesion, but may not tolerate extensive surgery, may have many co morbidities, may be prone to complications.
* Patients in whom surgery or radiation therapy may be impractical
* Primary lesions may be acceptable for enrollment
* Within normal limit hematopoietic capacity, hepatic and renal function. Values outside those limits may be allowed at the digression of the PI, if they are determined as not clinically significant
* Male patients must use condoms at all times, even after a vasectomy, during sexual intercourse with female partners of reproductive potential during treatment with vismodegib and for 3 months after the last dose to avoid exposing a pregnant partner and unborn fetus to vismodegib
* Male patients must agree not to donate sperm during the study and for 3 months after discontinuation of vismodegib
* Agreement not to donate blood or blood products during the study and for 7 months after discontinuation of vismodegib.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial.
* Ability to understand and the willingness to sign a written informed consent document in English

Exclusion Criteria:

* Women of childbearing potential
* Basal cell carcinomas of aggressive subtypes (infiltrative, morpheaform, micronodular)
* Any BCC that may require Mohs surgery for definitive control
* Subjects with porphyria's or known hypersensitivity to porphyrins
* Subjects with known photosensitivity diseases
* Subjects previously treated with a systemic photosensitizer within 4 months of screening date
* Subjects who desire to get pregnant a female of childbearing potential within the next 1.5 years
* Uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Life expectancy less than one year
* Inability or unwillingness to swallow capsules
* Have a history of alcohol of substance abuse, unless in full remission for greater than 6 months prior to the screening visit (Day 0) when the consent form is signed.
* Known to be infected with human immunodeficiency virus (HIV), hepatitis B or hepatitis C viruses.
* Currently receiving vismodegib, biologics or chemotherapy
* Currently undergoing treatment with photodynamic therapy, topical chemotherapy agents including Imiquimod, fluorouracil, Ingenol mebutate (picato) to the selected treatment lesion sites.
* Subjects who have Gorlins syndrome
* Subjects who have received any type of solid organ transplant
* Subjects taking immunosuppressive medications at the screening visit.
* Participation in other study using an investigational or experimental therapy or procedure within 4 weeks or 5 half-lives (whichever is longer) before the screening visit and/or during study participation. Subjects cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects unable or unwilling to comply with the study visit schedule and requirements of the study
* Subjects unable to speak and read the English language
* A subject who, in the opinion of the sponsor-investigator will be uncooperative or unable to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
The number of participants with treatment related adverse events as assessed by the CTCAE v4.0 | 2 years
  The proportion of evaluable study participants who had a grade 3 or higher adverse event (AE) or any serious adverse event that's determined to be at least possibly or probably related to study treatment, or any AE which is at least possibly or probably related to study treatment that causes permanent study discontinuation.

SECONDARY OUTCOMES:
The number of participants with overall response rate | 2 years
  To evaluate the overall response rate (ORR) to the combination therapy in patients with multiple BCCs. ORR is defined as the proportion of evaluable study subjects who has complete or partial response to the study treatment.
  Complete response (CR): Disappearance of all target lesions Partial response (PR): At least a 30% decrease in the sum of the diameters of target lesion, taking as reference the baseline sum diameters.
The number of participants wtih progressive disease or stable disease | 2 years
  The proportion of evaluable subjects with progressive disease (PD), and the proportion of evaluable subjects with stable disease (SD). Progressive Disease (PD): At least a 20% increase in the sum of the diameter of target lesions, taking as references the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of one or more new lesions is also considered progression.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or sufficient increase to qualify for PD, taking as reference the smallest sum diameter while on study. Subjects having a documented response with no confirmation of the response will be listed with stable disease.
The number of patients with complete histological clearance | 2 years
  Complete histological clearance (CHC): Negative for BCC on punch biopsy at the end of the follow up visits.
Overall treatment related pain during PDT assessed with the 11 point visual analogue scale (VAS) . | 2 years
  Pain scores (VAS) of each patientwill be recorded at three time points (beginning, midway and end of PDT session). The mean score (±) SD of the study population will be calculated at each time point. Mean pain scores of study population will be compared with each other. In addition Mean Difference of pain scores before and after PDT of each patient will be calculated and an average (sum) of mean difference values of all patients will be measured
Overall cosmetic scores on a scale of 1-5. | 2 years
  Cosmesis will be evaluated by the investigator at the end of treatment and be rated as 1. Poor (hypertrophic scarring, significant hypo/hyper pigmentation), 2. Fair (flat scar,moderate pigmentation changes ) 3 .Good (mild pigmentation changes and scar changes) 4. Excellent (min to no pigmentation changes) 5. Still healing.The cosmetic scores will be recorded after all treatments, and tabulated for each lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Mariette Marsh, Study Chair — University of Arizona Human Subjects Protection Program
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided